CLINICAL TRIAL: NCT02000362
Title: An Open-labelled, Multi Center, Comparative Phase I/IIa Clinical Trial to Evaluate the Efficacy and Safety of FURESTEM-CD Inj. in Patients With Moderately Active Crohn's Disease
Brief Title: Safety and Efficacy of FURESTEM-CD Inj. in Patients With Moderately Active Crohn's Disease(CD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSTHD_FURESTEM-CD
Record Dates: First submitted 2013-11-07; First posted 2013-12-04 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2016-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Stem cell; Cell therapy; Auto-immune disease; furestem; CD; inflammatory bowel disease; MSCs; Mesenchymal Stem Cells; hUCB-MSC; UCB-MSC; Umbilical cord Blood
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): cohort 1. 5.0 x 10^7 stem cells after registration
  cohort 2. 1.0 x 10^8 stem cells after registration
  Interventions: Biological: Stem cells

INTERVENTIONS:
Biological: Stem cells
  Other Names: FURESTEM-CD Inj.

SUMMARY:
The purpose of phase I clinical trial is to evaluate safety and efficacy in subjects with moderately active Crohn's disease after injection for 28days.

The purpose of phase IIa clinical trial is to determine therapeutic safety and efficacy of FURESTEM-CD Inj. which is based on Crohn's disease activity index(CDAI)<150 after injection.

DETAILED DESCRIPTION:
Crohn's disease is mysterious chronic inflammatory bowel disease. It usually happen in the young age and last forever. It is not yet clearly known the origin of crohn's disease. However, crohn's disease therapy is getting developed by using immunosuppressant and TNF-alpha inhibitor. Nonetheless, some patients still don't react to TNF-alpha inhibitor which is most effective treatment. Also, Even though some other patients reacted to the treatment at first, the effect of treatment decreases over time. Plus, long-term use of TNF-alpha inhibitor can lead to complication of infection and occurrence of malignant tumor like lymphoma. Recently, treatment of intractable crohn's disease is attempted by using stem cell. Especially, Mesenchymal stem cell is well-known for immunosuppression, anti-inflammatory ability and cell differentiation ability to various lineage cell as non hematopoietic stromal cell.

When the body get infected by the pathogens, innate immune response operate as the primary defence mechanism. at this time, there are some receptors reacting first such as TLR(toll-like receptor) and NLR(nucleotide-binding oligomerization domain) which is located in the cytoplasm of a cell. It is reported that the activities of TLR which is expressed by Mesenchymal stem cells play an important roles about immunomodulatory ability of Mesenchymal stem cells. Furthermore, human Umbilical Cord Blood derived-Universal Stem Cells( hUCB-USCs) manifest TLR and NLR of Mesenchymal Stem cells at the same time. when those receptors become activation, it maximize ability of immunomodulatory. Therefore, hUCB-USCs can be utilized to cure intractable autoimmune disease like Crohn's disease. Further, It has huge possibility as cell therapy products for autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

1. of either gender, aged≥19 and ≤70 years
2. subjects who is diagnosed with Crohn's disease after considering all the factors below.

   1. histological or pathological Diagnostic opinion
   2. colonoscopic Diagnostic opinion
   3. radiologic and hematological Diagnostic opinion
3. subjects who is included in two criteria below and come under CDAI 220-450 during screening period.

   1. CRP>0.3mg/dL during screening period
   2. more than 3 nonanastomotic ulcers which is included in Crohn's disease as a result of colonoscopy on screening period(each diameter of ulcers needs to exceed 0.5cm)
4. range of Crohn's disease : an affection of ileum, an affection of large intestine, an affection of ileum and large intestine at once.
5. subjects who suffer from extensive colitis during more than 8 years or limited colitis during more than 12 years need to have evidence that there are no large intestine ulcers by surveillance colonoscopy on screening visit.
6. subjects who are included in two criteria about drug treatment of Crohn's disease like below.

   1. subjects who fail the existing treatment and come under more than 1 criterion as below.

      * subjects who continuously administer Corticosteroid or immunosuppressant (AZA, Methotrexate, 6-MP)
      * subjects who have history of improper response or intolerance about Corticosteroid or immunosuppressant (AZA, Methotrexate, 6-MP)
      * subjects who are dependent Corticosteroid or have history of Corticosteroid dependence.
   2. subjects who have history of improper response or intolerance about anti-TNF treatment as below.

      * Infliximab
      * Adalimumab
      * Certolizumab pegol
7. subjects who satisfy those clinical examination value below during screening period.

   * Hemoglobin ≥ 8.0g/dL
   * WBC ≥ 3,000/μL
   * Lymphocyte ≥ 500/μL
   * 100,000/μL ≤ Platelet ≤ 1,200,000/μL
   * AST and ALT ≤ 3 x the upper limit of normal
   * ALP ≤ 3 x the upper limit of normal
   * Serum creatinine ≤ the upper limit of normal
   * Serum albumin ≥ 2.0g/dL
   * PT ≤ the upper limit of normal
   * aPTT ≤ the upper limit of normal
8. subjects who agree with those use of contraceptive method during clinical trial period.

   1. woman : subjects who is applicable to more than 1 case below.

      * subjects who is postmenopausal for more than 1 years before screening visit.
      * surgically sterility.
      * If subjects are biological clock, subjects need to agree with prohibition on having sex with man or usage of more than 2 effective contraception from sign of informed consent form until end of the clinical study.
   2. man : even surgically sterility(for example, getting a vasectomy), in case of satisfy those conditions below.

      * subjects who agree with prohibition on having sex with woman or usage of effective barrier contraception from sign of informed consent form until end of the clinical study.
9. subjects who understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Exclusion Criteria of gastrointestinal tract

   1. Crohn's disease which is invaded only proximal ileum.
   2. the evidence of an intra-abdominal abscess during screening period.
   3. the evidence of an abscess around the anus during screening period.
   4. conditions of subtotal colectomy or total colectomy.
   5. short bowel syndrome.
   6. subjects who conduct elemental diet, tube feeding or parenteral nutrition within 3 weeks before registration.
   7. subjects who have ileostomy or colostomy.
   8. subjects who remove existing seton before screening period.
   9. fixed bowel stricture which has symptoms.
   10. In case that the PI anticipate that subjects need to get a surgical intestinal tract surgery caused by Crohn's disease.
   11. non-removal of large intestine adenoma.
   12. chronic inflammation-associated dysplasia.
2. Exclusion Criteria of drugs

   1. in case subjects administered more than one drug within 4 weeks before enrollment.

      * Cyclosporine, tacrolimus, thalidomide
      * Adalimumab
      * Intravenous adrenocortical steroid
   2. in case subjects administered more than one drug within 10 weeks before enrollment.

      - Infliximab
      * Cetolizumab pegol
      * All kinds of biologicals
   3. in case subjects administered 5-ASA or Corticosteroid local treatment(a suppository or enema) within 2 weeks before enrollment.
   4. in case concomitant drug use for CD treatment cannot observe stable dosage during clinical study period or specified period like below.

      * use of oral 5-ASA compound at least 4 weeks before enrollment
      * use of oral Corticosteroid (prednisolone ≤ 20mg/day or budesonide ≤9mg/day) at least 2 weeks before enrollment
      * use of antibiotics for CD treatment at least 2 weeks before enrollment. (ex. metronidazole)
      * use of immunosuppressant at least 4 weeks before enrollment.
3. Exclusion Criteria of infectious disease

   1. acute or chronic hepatitis like below(typeA, typeB, typeC).

      * IgM anti-HAV positive
      * HBs-Ag, IgM anti-HBc, IgG anti-HBc positive. (It is possible to enroll the clinical study when a subject is anti-HBs Ab positive, given that the subject is both HBs-Ag and IgM anti-HBc negative or IgG anti-HBc positive.)
      * HCV-Ab positive
   2. tuberculosis

      * status present active tuberculosis
      * latent tuberculosis : subjects who is applicable to more than 1 case below.

        * QuantiFERON TB-GOLD positive or 2times continuous indeterminate within 4weeks before registration.
        * more than 10mm in tuberculin skin test within 3 months before registration.(when subjects got injected prednisolone more than 15mg per day, limited tuberculin skin test value is 5mm)
        * In case of observation of pulmonary tuberculosis cicatrix through X-Ray within 3months before registration.
   3. All kinds of Congenital or Acquired Immunodeficiency Syndrome.
   4. all kinds of live vaccine inoculation except influenza vaccine within 4weeks before registration.
   5. Clinically Significant infection with in 4weeks before screening visit or during screening visit.(pneumonia, pyelonephritis, Infection of Clostridium difficile etc.)
4. General exclusion Criteria a. subjects who experienced stem cell therapy. b. History of a malignant tumor except as noted below.

   * properly cured non-metastatic basal cell skin cancer
   * properly cured pinacocyte skin cancer which is not recurred at least 1 year before registration.
   * properly cured carcinoma in situ of uterine cervix which has not recurred at least 3 years before registration.

     c. malignant tumor which is not cured yet. d. subjects who are breast-feeding. e. unstable and not regulated disease(associated with cardiovascular, lung, liver, kidney, gastrointestinal tract, urogenital organs, hematologic, immune, endocrine/metabolism, etc.) which has possibility to hamper safety of subjects or cause confusion in clinical study.

     f. subjects who got general anesthesia surgery within 4weeks before registration or subjects who anticipated necessity of general anesthesia surgery during clinical study.

     g. major neurological history including stroke, multiple sclerosis, encephaloma, neurological degenerative disease.

     h. history of hypersensitive reaction about MR contrast medium. I. history of addictive drugs or alcohol with 1 years. j. active psychiatric problem which can hamper participation of clinical study. k. all kinds of problems which has possibility to hamper participation of study visit and observance of study procedure.

     l. Any other condition which the PI judges would make subject unsuitable for study participation.

     m. subjects who got injected other investigational product within 4 weeks or at present.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events, Ratio of patients who is applicable to CDAI<150 | 4 weeks follow-up after treatment, 12 weeks follow-up after treatment
  on phase 1, Phase 2a

SECONDARY OUTCOMES:
the ratio of patients who reduce CDAI over 70 as contrasted with baseline value | 12 weeks follow-up after treatment
  on phase 2a
a variation of CRP value as contrasted with baseline | 12 weeks follow-up after treatment
  on phase 2a
a variation of MR enterographic score as contrasted with baseline | 12 weeks follow-up after treatment
  on phase 2a
a variation of fecal calprotectin as contrasted with baseline | 12 weeks follow-up after treatment
  on phase 2a
a variation of IBDQ score as contrasted with baseline | 12 weeks follow-up after treatment
  on phase 2a
a variation of SF-36 score as contrasted with baseline | 12 weeks follow-up after treatment
  on phase 2a
reduction of the number of draining fistula | 12 weeks follow-up after treatment
  on phase 2a
all kinds of adverse effects which occur during the clinical study | 12 weeks follow-up after treatment
  on phase 2a

CONTACTS AND LOCATIONS:
Overall Officials: Suk-kyun Yang, Principal Investigator — Asan Medical Center
Locations (7):
- South Korea (7):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Seoul National Universtiy Bundang Hospital, Seongnam-si
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Soeul National University Hospital, Soeul
  - The Catholic University of Korea, St. Vincent'S Hospital., Suwon